CLINICAL TRIAL: NCT00880360
Title: A Phase II Trial of Intravenous Ontak to Treat Epithelial Ovarian Cancer FIGO Stage III or Stage IV, or Extraovarian Peritoneal Carcinoma, of Fallopian Tube Carcinoma Failing or Ineligible for First-Line Therapy
Brief Title: A Trial of Intravenous Denileukin Diftitox in Stage III or IV Ovarian Cancer
Acronym: ONTAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20070042H; OCR 07-04 (Other: UTHSCSA); NCT00238186 (obsolete NCT alias)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2013-01

CONDITIONS: Epithelial Ovarian Cancer; Extraovarian Peritoneal Cancer; Fallopian Tube Carcinoma
Keywords: Epithelial Ovarian Cancer; FIGO (International Fed of Gyn and Ob)Stage III or Stage IV; Extraovarian Peritoneal Cancer; Fallopian Tube Carcinoma Failing
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ontak (Experimental): Administration of Ontak IV for treatment of epithelial ovarian cancer
  Interventions: Drug: Ontak

INTERVENTIONS:
Drug: Ontak — Patients will be treated with Ontak at 12 µg/kg monthly as long as they meet response criteria.
  Other Names: Denileukin Diftitox

SUMMARY:
This study tests whether denileukin diftitox will deplete regulatory T cells, boost tumor-specific immunity and treat epithelial ovarian cancer in patients who have failed, or who are ineligible for front line therapy.

DETAILED DESCRIPTION:
This is a non-randomized, single-arm, Phase II trial. Selected patients with advanced-stage epithelial ovarian cancers who have no reasonable chance of cure using standard regimens, or who will not receive such regimens (due to contraindication or intolerance) are eligible. Patients will be treated with Ontak at 12 µg/kg monthly as long as they meet response criteria.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Not on Immune modulating drugs
* Life expectancy less than 6 months

Exclusion Criteria:

* Unable to tolerate phlebotomy
* Germ cell or stromal cell cancers of the ovaries
* Active autoimmune disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Curiel, MD, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- CTRC at UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ontak: Ontak : Patients will be treated with Ontak at 12 µg/kg monthly as long as they meet response criteria.
Period: Overall Study
Arm/Group | Ontak
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ontak
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Clinical Response
Description: Assess the efficacy of Ontak to treat selected advanced-stage ovarian epithelial cancers measured by clinical response rate, disease-free progression, and overall survival.
Time Frame: 2 years
Population: Measurements performed by RECIST criteria and response reported as a percent. 56 subjects needed to be recruited to the study to determine efficacy. Analysis was on an intent to treat basis.
Measure: Number; unit: participants
Arm/Group | Ontak
Number analyzed (Participants) | 19
participants | 19

2. Secondary Outcome: Toxicity
Description: Determine any toxicity associated with Ontak treatment in these patients.
Time Frame: 3 years
Population: N/A data were not collected
Arm/Group | Ontak
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ontak
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No